CLINICAL TRIAL: NCT02039596
Title: Nutritional Metabolomics: the Search for Dietary Exposure Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Nutritional Metabolomics AIKN; 2011-20497-84904-38 (Other Grant/Funding Number: The Swedish Research Council)
Record Dates: First submitted 2013-12-17; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Nutrition Disorders; Metabolic Disorders
MeSH Terms: conditions — Nutrition Disorders; Metabolic Diseases | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- vegetarian breakfast (Experimental): Diet: Vegetarian food items
  Interventions: Other: Diet
- Swedish Breakfast (Experimental): Diet: Swedish food items
  Interventions: Other: Diet
- English breakfast (Experimental): Diet: English food items
  Interventions: Other: Diet
- Lacto-vegetarian breakfast (Experimental): Diet: Lacto-vegetarian food items
  Interventions: Other: Diet
- Swedish omnivore breakfast (Experimental): Diet: Swedish breakfast with meat items
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet

SUMMARY:
In the post-genomic era, a major challenge for health research is to understand the complex interactions among genetic, environmental and lifestyle factors including dietary intake. Unfortunately, such initiatives are hampered by the lack of accurate dietary intake assessment methods for large studies. The newly emerging field of metabolomics offers unique possibilities to characterize individual food intake, dietary patterns and effects of dietary intervention in large studies. The investigators propose to develop a platform to detect broad metabolomic responses to food intake in controlled trials as well as to use targeted metabolomics approaches to characterize dietary intake in longitudinal studies. Our laboratory has a long history of developing methodology for assessing nutritional status and effects of diet on metabolism. Here, the investigators team up with the Sahlgrenska Academy Core Facility and the Swedish NMR Centre at the University of Gothenburg, that offer modern metabolomics equipment and competence in bioinformatics, and use this in the context of nutrition research. To their knowledge, the investigators are among the first groups in the country to develop skills in metabolomics to assess dietary intake and effects of nutrition on metabolism, and probably the first to use two complementary platforms with both mass-spectrometry and nuclear magnetic spectroscopy. Hence, our methodological results should be useful to nutritional scientists nationally as well as internationally.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5-30.0
* Age 18-65 years old

Exclusion Criteria:

* Medications or tobacco use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Acute metabolomic response | Directly after ingestion of test meal
  The acute metabolomic response (ie all metabolites) to a test meal will be analyzed using both nuclear magnetic resonance (NMR) and mass spectrometry (MS) techniques. Patterns of metabolites will be evaluated with statistical techniques, ie discriminant analysis and principal component analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anna K Winkvist, PhD, Principal Investigator — Univ of Gothenburg, Sweden; Lars H Ellegard, PhD, MD, Study Chair — Univ of Gothenburg; Helen M Lindqvist, PhD, Study Director — Univ of Gothenburg
Locations (1):
- Dept Internal Medicine and Clinical Nutrition, Univ of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Radjursoga M, Lindqvist HM, Pedersen A, Karlsson GB, Malmodin D, Brunius C, Ellegard L, Winkvist A. The 1H NMR serum metabolomics response to a two meal challenge: a cross-over dietary intervention study in healthy human volunteers. Nutr J. 2019 Apr 8;18(1):25. doi: 10.1186/s12937-019-0446-2. PMID 30961592